CLINICAL TRIAL: NCT04237519
Title: StayFitLonger. Preventive Effects of a Combination of Non-drug Interventions (Physical, Cognitive and Social) in Healthy Elderly Subjects: Multicentre Randomised Controlled Trial.
Brief Title: The StayFitLonger Study: an Innovative Computerized Home-based Training to Foster Independent Life at Home
Acronym: SFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: HES-SO Valais-Wallis (Other); Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); Haute-Ecole Arc (Unknown); Mindmaze SA (Industry); Université Catholique de Louvain (Other); Active and Assisted Living Programme (Unknown); BRUSANO (Unknown); Pro-Senectute Vaud (Unknown)
Responsible Party: Principal Investigator, Jean-François Démonet, Professor, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: aal-call-2017-068
Record Dates: First submitted 2020-01-13; First posted 2020-01-23 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Decline Prevention in Robust Older Adults; Cognitive Decline Prevention in Pre-frail Older Adults; Physical Decline Prevention in Robust Older Adults; Physical Decline Prevention in Pre-frail Older Adults
Keywords: Multimodal intervention; Cognitive training; Physical training; Social interactions; Prevention; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel-group (intervention A vs B), multicentric randomized control trial (RCT). A stratification will separate robust from pre-frail healthy older adults in each intervention.
  Note that the study is combined with a further 6-month observational study to test adherence, user experience and acceptability in all participants.
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors are blind to the hypotheses and to participants' assignment as they only have access to the testing sessions. Participants are asked not to mention elements of their training program to assessors . Would such circumstance occur, it will be reported but this should have minimal effect on integrity as the assessors are blind to the hypotheses.
  Team members responsible of the statistical analyses are blind to the training assignment as they only have access to anonymized data set and have no access to neither participants' assignment nor the randomization list.
  At each study site, study coordinators and trainers responsible for the introductory and refresher courses, and supervision of participants during the home-based training are not blind.
  Participants are aware that the trial has two different training conditions that are compared to each other and that they are randomly allocated to one of them. However, they are not informed of the study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFL training (Experimental): Practice recommendation 3 times per week:
  * Physical exercises: between 30 to 45 minutes that can be split during the day (e.g. 2x15 or 20 minutes, or 3x10 or 15 minutes during the same day).
  * Cognitive exercises: minimum of 15 min.
  Interventions: Behavioral: SFL training
- Active control training (Active Comparator): Practice recommendation 3 times per week:
  * Physical exercises: between 30 to 45 minutes that can be split during the day (e.g. 2x15 or 20 minutes, or 3x10 or 15 minutes during the same day).
  * Cognitive exercises: minimum of 15 min.
  Interventions: Behavioral: Active controlled training

INTERVENTIONS:
Behavioral: SFL training — The SFL training program comprises:
  * Physical exercises: 50 video exercises to improve balance, muscle strength and physical capabilities in older adults;
  * Cognitive exercises: Four ludic activities targeting problem solving (4 Images/ 1 word), memory (Quiz and Recall me), speed processing and divided attention (Attention!).
  In addition, the SFL program includes a series of unique components:
  * Chat rooms: to share views about topics of interest and tips for common real-life problems;
  * Psycho-education content: to improve self-management and promoting cognitive transfer though 22 different topics (provide recommendations usually given in psychotherapy sessions);
  * Virtual coach: to guide participants along the proposed exercises by giving them instructions, reminding them regularly to practice a variety of available activities repeatedly, providing appropriate and timely feedback on participant's performances and rewarding assiduity, perseverance and performance.
  Arms: SFL training
Behavioral: Active controlled training — The active control training program is structured in the same manner as the SFL training program and will also offer different physical and cognitive activities:
  * Physical exercises: 12 different exercises trains upper and lower extremity strength, mobility and balance offered through a computerized version of a health insurance company physical training program;
  * Cognitive activities: Four commercially available leisure activities (Sudoku. Cross Words, Pac-Man and Countdown activities) that are appreciated by older adults but do not teach cognitive strategies and are were not designed to improve cognition per se.
  No chat room, psycho-educational content or virtual coach were included in the active control training program.
  Arms: Active control training

SUMMARY:
Multimodal training, including physical and cognitive activities, has been associated with a reduction in age-related physical and cognitive decline. Therefore, combining these activities into a home-based computerized training program may represent a powerful approach to foster independent life at home. The StayFitLonger study is a 6-month multi-site randomized controlled, double-blind trial, which tests the efficacy of a home-based computerized intervention that combines physical and cognitive exercises through virtual coaching to enhance motivation.

In Switzerland, Canada and Belgium, a total of 128 older participants will be recruited and randomly assigned to one of two physical and cognitive home-based interventions for 6 months: StayFitLonger or active control training. The StayFitLonger intervention provides physical and cognitive training exercises, feedback and instructions through a virtual coach to optimize motivation. It also offers social and psycho-educational contents. Monthly supervision (home-visits and phone calls) will be provided during this 6-month intervention. Outcomes will be measured at baseline, and after 6 months of training.

This study will demonstrate the feasibility, sustainability and efficacy of a home-based multi-domain intervention program allowing further development and possible commercialization of a scientifically validated training program to slow down cognitive and physical decline.

DETAILED DESCRIPTION:
Finding ways to improve and maintain functional abilities and quality of life in older people has become a worldwide priority. It is well recognized that reduced engagement in physical, cognitive and social activities has negative influence on the health of older adults. This leads to more vulnerabilities both physically and cognitively. Sedentary behaviors can ultimately induce physical frailty, defined as a state of high vulnerability with accumulation of adverse health outcomes. Fear of falling and/or unsteady gait are common factors of physical frailty. Moreover, falls are particularly common in older adults. In addition to mobility limitation and falls, cognitive decline has been identified as a major cause of disability and dependency in older populations.

Through non-pharmacological interventions focusing on alterable lifestyle factors, experts believe in the possibility to protect older people from the deleterious effects of physical and brain aging that can lead to dementia. In other words, keeping a healthy mind in a healthy body might be the gold standard for healthy aging. Several studies have shown that physical activity, through aerobic, gait and strength training, induces many beneficial effects including improvement of general health, cognition and quality of life. In addition, a growing number of cognitive interventions have been conducted in healthy seniors and older adults with mild cognitive impairment (MCI) and results show improved cognition and delayed cognitive decline. As well, cognitive deficits, mainly in executive functions, have been associated with an increase number of falls and abnormal gait among others.

Improvement of these physical functions was observed in response to cognitive interventions. Because aging is complex and different interventions are likely to potentiate their effects, an increasing number of studies have reported on combined interventions targeting two or more modifiable factors. However, accessibility to these interventions remain a major challenge because older adults may not have access to specialized expertise and resources.

The use of a computerized system to deliver lifestyle interventions have several advantages: it can be used to support home-based training, reducing costs and increasing access; training can be self-paced and last over practically a unlimited time; it allows providing immediate feedback; it offers potential for scaling up for wider use if efficacy is proven; it provides an excellent interface for active control interventions. Surprisingly, whereas many studies assessed computerized cognitive training programs, only a few have used home-based interventions which combine cognitive training with physical activity and, to our knowledge, only one study used computerized tasks for both physical and cognitive training in healthy older adults.

The StayFitLonger study was designed to test efficacy of a home-based computerized training program targeted at older adults, which combine physical exercises and cognitive training. The main goal of the program is to improve physical health and prevent frailty through an innovative approach using videos of 50 physical exercises focusing on gait and strength, which could be easily implemented in older adults (Test-and-Exercise home-based program). The program was also designed to enhance cognitive functions through a series of activities in form of serious games. These activities train executive control through dual-task exercises that was found to increase divided attention and frontal lobe function general knowledge learning and problem solving training. Other features of the program that are unique include: 1) Prospective memory exercises embedded in the physical exercises; 2) Social interactions whereby participants can create and share with other participants their learning material and can chat with their peers about topics of interest and find solutions to common real-life problems; 3) Psycho-educational content on cognition, physical health, nutrition and on ways to apply newly learned strategies in real life to empower participants and promoting self-management; 4) A virtual coach aimed to improve adherence by guiding participants, reminding them to use the program regularly, and providing feedback and rewards through a system of virtual credits; 5) Possibility to personalize the application settings to tailor the environment to the participant's tastes and wishes; 6) Wearable motion sensors used during physical exercises for movement detection as a game input and for providing measurements on mobility for a better characterization of the potential benefits of the program.

The StayFitLonger study will test the effect of the training on key outcomes using a double-blind, parallel-group, randomised control trial (RCT) over 6 months. The primary objective is to assess whether the 6-month StayFitLonger programme leads to better performance than those observed following the active control condition on the Timed-Up & Go (TUG), a functional physical task, which is associated with lower-body strength and balance. The efficacy study also includes a few secondary objectives. One is to assess whether the StayFitLonger programme improves other physical capabilities as well as cognitive performances and scores of affective variables (e.g., mood, fear of falling), and psycho-social domains (e.g., quality of life, daily living activities, participant's expectation). In addition, the study will also assess whether a similar gain is found in robust vs pre-frail seniors.

In Switzerland, Canada and Belgium, a total of 128 older participants will be recruited. Following the initial eligibility screening, participants will be randomized to one of two home-based computerized intervention conditions, the StayFitLonger training program (experimental) or the active control training program . Enrolled participants will be evaluated at two time points: at baseline (T0) and after 6 months of training (T1, end of the RCT). The training will take place at home for 6 months. Prior to the start of the training and within a month following T0 assessment, introductory courses in groups of a maximum of 6 people will take place to introduce the features of the program and describe the different physical and cognitive exercises. Participants will be supervised through home visits and monthly phone calls to ensure a good use of the program in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Fluent french speaker adults
* Retired, living at home and having a wireless Internet connection in their house;
* Independent for all daily activities (optimal score to the 4-IADL);
* Open to the use of new technologies and electronic tablets;
* Interested in exercising to stay fit;
* Able to walk without a walking aid (e.g. wheelchair, sticks, walker, etc.);
* Available to commit themselves for the time period during which the study takes place;
* No vision deficits that would prevent them to read information on a tablet;
* No current neurological or psychiatric diagnosis (e.g. Parkinson's disease).

Exclusion Criteria:

* MoCA score < 26;
* score ≥ 3 on the Fried's frailty index (Fried et al., 2001)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Timed-Up & Go Test (TUG) | T0 (baseline)
  To measure lower extremity function, mobility and risk of falls
Timed-Up & Go Test (TUG) | T1 (six months following T0)
  To measure lower extremity function, mobility and risk of falls

SECONDARY OUTCOMES:
Physical domain: Twenty-meter walking test | T0 (baseline)
  To measure gait speed in sec.
Physical domain: Twenty-meter walking test | T1 (six months following T0)
  To measure gait speed in sec.
Physical domain: Five Time Sit to Stand Test (FTSTS) | T0 (baseline)
  To measure lower extremity strength in sec
Physical domain: Five Time Sit to Stand Test (FTSTS) | T1 (six months following T0)
  To measure lower extremity strength in sec
Physical domain: Four Stage Balance Test (FSBT) | T0 (baseline)
  To measure balance. A total score of 4 is obtained when a participant performs successfully 4 positions (parallel, semi-tandem and tandem). The test is stopped when a participant fails at holding a given position for at least 10 sec.
Physical domain: Four Stage Balance Test (FSBT) | T1 (six months following T0)
  To measure balance. A total score of 4 is obtained when a participant performs successfully 4 positions (parallel, semi-tandem and tandem). The test is stopped when a participant fails at holding a given position for at least 10 sec.
Physical domain: motion sensors measures | T0 (baseline)
  During TUG and 20-m walking test, motion sensors will provide measures on: walking speed, variability in gait, stance phase, foot-flat phase, double support, stride velocity, maximal swing speed, turning angle and variability in toe clearance.
Physical domain: motion sensors measures | T1 (six months following T0)
  During TUG and 20-m walking test, motion sensors will provide measures on: walking speed, variability in gait, stance phase, foot-flat phase, double support, stride velocity, maximal swing speed, turning angle and variability in toe clearance.
Cognitive domain: Global cognition composite score | T0 (baseline)
  This score is the ZAVEN composite score computed by averaging z-scores from:
  * Total recall of the California Verbal Learning Test (CVLT) and delayed recall of the WMS-IV Logical Memory to measure episodic memory;
  * WAIS-IV Digit Symbol substitution Test (DSST) to measure complex attention;
  * Verbal fluency (VF) to measure executive functions.
Cognitive domain: Global cognition composite score | T1 (six months following T0)
  This score is the ZAVEN composite score computed by averaging z-scores from:
  * Total recall of the California Verbal Learning Test (CVLT) and delayed recall of the WMS-IV Logical Memory to measure episodic memory;
  * WAIS-IV Digit Symbol substitution Test (DSST) to measure complex attention;
  * Verbal fluency (VF) to measure executive functions.
Cognitive domain: Memory composite score | T0 (baseline)
  This score is computed by averaging z-scores from:
  * Delayed recall of the CVLT;
  * Delayed recall of the WMS-IV Logical Memory Test.
Cognitive domain: Memory composite score | T1 (six months following T0)
  This score is computed by averaging z-scores from:
  * Delayed recall of the CVLT;
  * Delayed recall of the WMS-IV Logical Memory Test.
Cognitive domain: Executive composite score | T0 (baseline)
  This score is computed by averaging z-scores from:
  * Verbal fluency (VF);
  * Trail Making Test (condition B - A; shifting - processing speed scores);
  * Victoria Stroop (high interference - naming conditions);
  * Divided attention subtest from the Test of Attention Performance 2.3.1 (number of total omissions (visual and auditory)).
Cognitive domain: Executive composite score | T1 (six months following T0)
  This score is computed by averaging z-scores from:
  * Verbal fluency (VF);
  * Trail Making Test (condition B - A; shifting - processing speed scores);
  * Victoria Stroop (high interference - naming conditions);
  * Divided attention subtest from the Test of Attention Performance 2.3.1 (number of total omissions (visual and auditory)).
Cognitive domain: Speed processing composite score | T0 (baseline)
  This score is computed by averaging z-scores from:
  * Trail Making Test (time on condition A);
  * DSST (number of correct symbols);
  * Victoria Stroop (time on naming condition).
Cognitive domain: Speed processing composite score | T1 (six months following T0)
  This score is computed by averaging z-scores from:
  * Trail Making Test (time on condition A);
  * DSST (number of correct symbols);
  * Victoria Stroop (time on naming condition).
Affective domain: Hospital Anxiety and Depression Scale (HADS) | T0 (baseline)
  To measure mood.
Affective domain: Hospital Anxiety and Depression Scale (HADS) | T1 (six months following T0)
  To measure mood.
Affective domain: Falls Efficacy Scale International (FES-I) | T0 (baseline)
  To measure fear of falling.
Affective domain: Falls Efficacy Scale International (FES-I) | T1 (six months following T0)
  To measure fear of falling.
Psycho-social domain: Older People Quality of Life questionnaire (OPQOL 35). | T0 (baseline)
  To measure quality of Life (QoL)
Psycho-social domain: Older People Quality of Life questionnaire (OPQOL 35). | T1 (six months following T0)
  To measure quality of Life (QoL)
Psycho-social domain: Cognitive Function Instrument (CFI) - | T0 (baseline)
  To measure subjective difficulties encountered in activities of daily living, related to cognitive functions
Psycho-social domain: Cognitive Function Instrument (CFI) - | T1 (six months following T0)
  To measure subjective difficulties encountered in activities of daily living, related to cognitive functions
Psycho-social domain: Everyday Cognition (E-Cog) | T0 (baseline)
  To measure subjective difficulties encountered in activities of daily living, related to cognitive functions
Psycho-social domain: Everyday Cognition (E-Cog) | T1 (six months following T0)
  To measure subjective difficulties encountered in activities of daily living, related to cognitive functions
Psycho-social domain: Ad-hoc questionnaire | T0 (baseline)
  To measure participant's expectation from the training program. The questionnaire is related to the efficacy of the program and its different components, the expectation (difficulty, agreeableness, motivation) and the quality of the introductory courses.
Psycho-social domain: Ad-hoc questionnaire | T1 (six months following T0)
  To measure participant's expectation from the training program. The questionnaire is related to the efficacy of the program and its different components, the expectation (difficulty, agreeableness, motivation) and the quality of the introductory courses.
Cognitive processes manipulated during training: ad-hoc computerized test | T0 (baseline)
  To measure divided attention trained during Attention! activity with an ad-hoc computerized test designed specifically for this multitasking activity and provided in the form of a serious game.
Cognitive processes manipulated during training: ad-hoc computerized test | T1 (six months following T0)
  To measure divided attention trained during Attention! activity with an ad-hoc computerized test designed specifically for this multitasking activity and provided in the form of a serious game.
Cognitive processes manipulated during training: Rivermead Behavioural Memory Test - Third edition (RBMT-3). | T0 (baseline)
  To measure prospective memory trained in the Quiz activity with two subtests ("belonging" and "appointment")
Cognitive processes manipulated during training: Rivermead Behavioural Memory Test - Third edition (RBMT-3). | T1 (six months following T0)
  To measure prospective memory trained in the Quiz activity with two subtests ("belonging" and "appointment")
Cognitive processes manipulated during training: Flexibility subtest from the Test battery for Attention Performance | T0 (baseline)
  To measure concept elaboration trained in the 4images/1 word activity with a "set shifting" computerized task
Cognitive processes manipulated during training: Flexibility subtest from the Test battery for Attention Performance | T1 (six months following T0)
  To measure concept elaboration trained in the 4images/1 word activity with a "set shifting" computerized task
Cognitive processes manipulated during training: Similitudes subtest from the WAIS-IV: | T0 (baseline)
  To measure concept elaboration trained in the 4images/1 word activity and assess verbal reasoning and the development of concepts.
Cognitive processes manipulated during training: Similitudes subtest from the WAIS-IV: | T1 (six months following T0)
  To measure concept elaboration trained in the 4images/1 word activity and assess verbal reasoning and the development of concepts.

OTHER OUTCOMES:
Effects of moderators on primary and secondary outcomes: Age | Age measured within a month prior to the start of the intervention
  To see the influence of age on primary and secondary outcomes using 2 age groups defined by the median
Effects of moderators on primary and secondary outcomes: Sex | Sex measured within a month prior to the start of the intervention
  To see the influence of sex on primary and secondary outcomes using 2 sex groups (male and female)
Effects of moderators on primary and secondary outcomes: Education | Education measured within a month prior to the start of the intervention
  To see the influence of education on primary and secondary outcomes using 2 education groups (less or more than 12 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Demonet, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Sylvie Belleville, PhD, Principal Investigator — Institut universitaire de gériatrie de Montréal - CIUSSS; Stefan Agrigoroaei, PhD, Principal Investigator — Université Catholique de Louvain
Locations (4):
- Belgium (2):
  - BRUSANO (ASBL - Association Sans But Lucratif), Brussels
  - Centre Public d'Action Sociale, Woluwe-Saint-Lambert
- Institut universitaire de gériatrie de Montréal - CIUSSS du Centre-Sud-de-l'Île-de-Montréal, Montreal, Quebec, Canada
- Centre Leenaards de la mémoire - Centre hospitalier universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Derived] Belleville S, Cuesta M, Bieler-Aeschlimann M, Giacomino K, Widmer A, Mittaz Hager AG, Perez-Marcos D, Cardin S, Boller B, Bier N, Aubertin-Leheudre M, Bherer L, Berryman N, Agrigoroaei S, Demonet JF. Pre-frail older adults show improved cognition with StayFitLonger computerized home-based training: a randomized controlled trial. Geroscience. 2023 Apr;45(2):811-822. doi: 10.1007/s11357-022-00674-5. Epub 2022 Oct 21. PMID 36266559
- [Derived] Belleville S, Cuesta M, Bieler-Aeschlimann M, Giacomino K, Widmer A, Mittaz Hager AG, Perez-Marcos D, Cardin S, Boller B, Bier N, Aubertin-Leheudre M, Bherer L, Berryman N, Agrigoroaei S, Demonet JF. Rationale and protocol of the StayFitLonger study: a multicentre trial to measure efficacy and adherence of a home-based computerised multidomain intervention in healthy older adults. BMC Geriatr. 2020 Aug 28;20(1):315. doi: 10.1186/s12877-020-01709-2. PMID 32859156